CLINICAL TRIAL: NCT04020081
Title: A Pilot Study to Evaluate the Effect of Yoga Exercises and Meditation on Lung Volume, Respiratory Impedance, 6-minute Walk Distance and Quality of Life in Chronic Obstructive Pulmonary Disease(COPD) Patients.
Brief Title: A Study to Evaluate the Effect of Yoga Exercises and Meditation on Lung Function and Quality of Life in COPD Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chest Research Foundation, India (Other)
Collaborators: Jupiter Hospital, India (Unknown)
Responsible Party: Principal Investigator, Dr.Sundeep S Salvi, Director, Chest Research Foundation, India
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRF/01/2017
Record Dates: First submitted 2019-06-03; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: COPD; Obstructive Pulmonary Disease
Keywords: Yoga; Meditation; COPD; Lung function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of yoga exercises in COPD patients after 12 weeks. (Experimental): Yoga group
  Interventions: Other: Yoga breathing exercises and Meditation
- COPD patients lung functions without yoga excercises. (No Intervention): Control group

INTERVENTIONS:
Other: Yoga breathing exercises and Meditation — 8 Breathing exercises.The first set of 6 exercises is of the Upper Lobe breathing (Upper and Middle Lobe of the Lungs) while 7th exercise is abdominal breathing,8th exercise is yogic breathing.
  6-steps Nirmal Dhyan (meditation).Step 1: Breath awareness,Step 2: Body awareness,Step 3: Thought awareness,Step 4: Refreshing awareness,Step 5: Gap awareness,Step 6: Expanding awareness.
  Arms: Effect of yoga exercises in COPD patients after 12 weeks.

SUMMARY:
The Investigator would like to study the effect of yoga exercises and meditation on lung volume, respiratory impedance, 6-minute walk distance and quality of life in COPD patients.

DETAILED DESCRIPTION:
Hypotheses : The Investigator hypothesized that Yoga exercises improve the lung function (i.e. decrease in the lung hyperinflation, air trapping and airway impedance) by stretching the lung tissue, strengthening the respiratory muscles and increasing the chest expansion. Yoga exercises help to increase exercise capacity. Meditation reduces anxiety and depression.

Research Question: Do yoga exercises and meditation help to reduce respiratory impedance, hyperinflation, air trapping and increase exercise capacity and improve quality of life in COPD patients compared to control arm?

Objectives: 1. To study the effect of yoga exercises and meditation on exercise capacity and quality of life in COPD patients after 4, 8 and 12-weeks of intervention.

2.To evaluate residual volume (RV), residual volume/ total lung volume RV/TLC, total lung capacity TLC,inspiratory capacity/total lung capacity IC/TLC, and respiratory impedance in COPD patients after 4, 8 and 12-weeks of yoga exercises and meditation practice.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who is willing to provide written informed consent.
2. Male or female COPD patients aged ≥30 and < 70 years.
3. Subjects who are willing to do yoga exercises.
4. Clinical diagnosis of COPD confirmed on spirometry. Pre and post bronchodilator ratio of forced expiratory volume in 1sec/ forced vital capacity (FEV1/FVC) should be less than 0.7.

Exclusion Criteria:

1. Active smoker.
2. Pregnant women or nursing mothers. (Urine pregnancy test will be performed.)
3. Those unable to perform spirometry and body plethysmography.
4. Participants having symptoms of active pulmonary Koch's (tuberculosis).
5. Contraindications for spirometry: Subject having any of the following contraindications for spirometry.

   History of the following a) Recent (within 1 month) myocardial infarction. b) Unstable heart condition c) Hemoptysis (blood in sputum on coughing) in recent past (1 month) or d) A recent (within last one month) eye, chest or abdominal surgery.
6. Contraindications for Body Plethysmography: Subject having any of the following contraindications for body plethysmography

   1. Mental confusion, muscular in coordination, body casts, or other conditions that prevent the subject from entering the plethysmograph cabinet or adequately performing the required maneuvers (i.e., panting against a closed shutter).
   2. History of Claustrophobia.
   3. Presence of devices or other conditions, such as continuous intravenous infusions with pumps or other equipment that will not fit into the plethysmograph, that should not be discontinued, or that might interfere with pressure changes (e.g., chest tube, trans tracheal O2 catheter, or ruptured eardrum).
7. Anyone who is on continuous oxygen therapy
8. Patients who are doing yoga or taking pulmonary rehabilitation from last 6 months.
9. History of thoracic cage abnormality, musculoskeletal abnormality, interstitial lung disease, epilepsy
10. Patients who are unable to perform yoga exercises.
11. Contraindications for 6 Minute walk test:

    1. Absolute Contraindications: Unstable angina during the previous month and myocardial infarction during the previous month.
    2. Relative Contraindications : Resting heart rate of more than 120, a systolic blood pressure of more than 180 mm Hg, and a diastolic blood pressure of more than 100 mm Hg.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
St.George's Respiratory Questionnaires (SGRQ) score for quality of life in numbers. | 3 Months
  Effect of Yoga Exercises and Meditation on SGRQ score after 12 week in COPD patients.
Exercise capacity 6 minute walk distance (6MWD) in meter. | 3 Months.
  Effect of Yoga Exercises and Meditation on 6 minute walk distance (6 MWD) after 12 week in COPD patients.

SECONDARY OUTCOMES:
RV/TLC in% | 3 Months
  Effect of Yoga Exercises and Meditation on lung function after 12 week in COPD patients.
TLC in liters | 3 Months
  Effect of Yoga Exercises and Meditation on lung function after 12 week in COPD patients.
Respiratory impedance in kpa/(L/s) | 3 Months
  Effect of Yoga Exercises and Meditation on lung function after 12 week in COPD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sundeep Salvi, MD, Principal Investigator — Director
Locations (1):
- Chest Research Foundation, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donesky-Cuenco D, Nguyen HQ, Paul S, Carrieri-Kohlman V. Yoga therapy decreases dyspnea-related distress and improves functional performance in people with chronic obstructive pulmonary disease: a pilot study. J Altern Complement Med. 2009 Mar;15(3):225-34. doi: 10.1089/acm.2008.0389. PMID 19249998
- [Background] Kaminsky DA, Guntupalli KK, Lippmann J, Burns SM, Brock MA, Skelly J, DeSarno M, Pecott-Grimm H, Mohsin A, LaRock-McMahon C, Warren P, Whitney MC, Hanania NA. Effect of Yoga Breathing (Pranayama) on Exercise Tolerance in Patients with Chronic Obstructive Pulmonary Disease: A Randomized, Controlled Trial. J Altern Complement Med. 2017 Sep;23(9):696-704. doi: 10.1089/acm.2017.0102. Epub 2017 Jul 17. PMID 28714735
- [Result] Liu XC, Pan L, Hu Q, Dong WP, Yan JH, Dong L. Effects of yoga training in patients with chronic obstructive pulmonary disease: a systematic review and meta-analysis. J Thorac Dis. 2014 Jun;6(6):795-802. doi: 10.3978/j.issn.2072-1439.2014.06.05. PMID 24977005